CLINICAL TRIAL: NCT02726633
Title: Evaluate the Utility of the ProLung China Test as Adjunctive to CT Scan in the Diagnosis of Lung Cancer
Brief Title: Evaluate the Utility of the ProLung China Test in the Diagnosis of Lung Cancer
Acronym: ProLung
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Alliance Against Lung Cancer (Other)
Responsible Party: Principal Investigator, Bai Chunxue, Chair, Chinese Alliance Against Lung Cancer
Other Study IDs: CAALC-004-Prolung
Record Dates: First submitted 2016-03-29; First posted 2016-04-04 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Solitary Pulmonary Nodule; Multiple Pulmonary Nodules
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A Study to evaluate the utility of the ProLung China Test as an adjunct to CT scan in the diagnosis of lung cancer.

DETAILED DESCRIPTION:
This Study will assess the stability of the ProLung China Test classification algorithm when used as an adjunct to CT scan. This Study will assess whether there are any potential safety concerns of the ProLung China Test when used to evaluate patients with a positive CT scan for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, age 18 to 80.
2. Subject has undergone CT scan of the lung(s) that indicates one or more nodules or lesions.
3. Subject's pulmonary nodule or lesion is greater than 4mm and smaller than 50mm. Size is determined by the largest nodule or lesion dimension identified from CT imaging.
4. Subject must be able to receive a ProLung China Test within 30 days of abnormal CT within 14 days prior to the tissue biopsy or surgical resection.

Exclusion Criteria:

1. Subject has an implanted electronic device in the chest. Subject receiving therapy for suspected chest infection such as fungal infection or tuberculosis.
2. Subject with diagnosed malignancy other than lung cancer who has 2 or more suspicious pulmonary nodules.
3. Subject has received an invasive medical or surgical procedure within the thoracic cavity within 30 days prior to the ProLung China Test or within the previous 14 days for a bronchoscopic procedure.
4. Subject presents with an anomalous physical or anatomical condition that precludes ProLung China Test measurement.
5. Subject will have undergone unusually strenuous exercise within 24 hours.
6. Subject who has significant systemic diseases such as uncontrolled diabetes, advanced heart failure, or a recent myocardial infarction, or other medical condition such as severe morbid obesity that in the judgment of the Principal Investigator would make him/her unsuitable for the Study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with pulmonary lesions suspicious for lung cancer
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Efficacy of the ProLung China Test | The ProLung China Test will be performed within 30 days of a CT Scan that identifies a lung lesion suspicious for lung cancer and evaluated once a patient diagnosis is obtained.
  Demonstrate safety and efficacy in the risk stratification of patients with pulmonary lesions identified by CT that are suspicious for lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Chunxue Bai, MD, Study Chair — Chinese Alliance Against Lung Cancer
Locations (3):
- China (3):
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Shanghai Dongfang Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided